CLINICAL TRIAL: NCT04056832
Title: Left Ventricular Reverse Remodeling in Aortic Valve Replacement With Single Strip Pericardium and Mechanical Valve: A Comparative Study
Brief Title: Left Ventricular Reverse Remodeling In Aortic Valve Replacement With Single Strip Pericardium Versus Mechanical Valve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 011; ETIKUI-1612576 (Other: Ethical Committee of Universitas Indonesia)
Record Dates: First submitted 2019-02-01; First posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Aortic Valve Stenosis; Aortic Stenosis; Valve Stenoses, Aortic; Aortic Valve Calcification
Keywords: Aortic Stenosis; Aortic Valve Replacement; Single Strip Pericardium; Autologous Pericardium; Mechanical Valve Replacement; Comparison of Left Ventricle Remodeling
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve, Calcification of

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Strip Pericardium (Experimental): Aortic Valve Replacement using single strip of patient's autologous pericardium
  Interventions: Procedure: Single Strip Pericardium
- Mechanical Prosthetic Valve (Active Comparator): Aortic Valve Replacement using mechanical prosthetic valve
  Interventions: Procedure: Mechanical Prosthetic Valve

INTERVENTIONS:
Procedure: Single Strip Pericardium — The anterior pericardium is taken in accordance with the measurements made using an aortic annulus sizer or Ismail sizer. The diameter of the annulus valve is converted to circumference of the aortic valve according as a measure of the length of the pericardium. Measurement of aortic commissure height is done by measuring the distance between the lowest point of the valve attachment to the highest point on the commissure as a measure of pericardium width. The pericardium is immersed in 0.6% glutaraldehyde solution for 10 minutes, then rinsed and soaked with saline solution 3 times for 6 minutes each. After the pericardium becomes firm it is cut to be a single strip according to the length and width in the previous measurement. It is then sutured to the aortic valve annulus.
  Other Names: Autologous Pericardium
  Arms: Single Strip Pericardium
Procedure: Mechanical Prosthetic Valve — Median incision is performed at the surgical site. Sternal retractor is placed at the sternum after median sternotomy being performed. Aortic valve is measured using aortic annulus sizer. Pledgeted suture is performed for the mattress. Sutures are performed to attach the mechanical prosthetic to the aortic annulus.
  Arms: Mechanical Prosthetic Valve

SUMMARY:
Aortic stenosis is a commonly found heart disease, which often leads to mortality and morbidity. Valve replacement using mechanical prosthetic valve will have an expensive cost especially in the Integrated Heart Center of Cipto Mangunkusumo Hospital, Jakarta, Indonesia. In addition to the expensive cost, patients who have mechanical prosthetic valve have an increased risk of infection of the prosthetic valve and developing thrombo-embolism thus have to consume a lifelong anticoagulant therapy that increase risk of bleeding. A surgical technique using autologous pericardium is an alternative to prosthetic valve replacement, one of which is a single pericardium strip technique that uses modified autologous pericardium technique from Ozaki et al and Duran et al.

The objective of this study is to investigate the outcome of aortic valve replacement with a single pericardium strip of autologous pericardium in patients with aortic stenosis.

This study will be conducted at the Integrated Heart Center of Cipto Mangunkusumo Hospital, Jakarta, Indonesia, by using quasi experimental type time series design. Subjects are patients with aortic stenosis who are candidates for valve replacement. Inclusion criteria is having low to moderate surgical risk (EuroScore II <5). The sampling method used in this study is non-probability consecutive sampling. This study will assess the outcome of the aortic valve replacement (valve hemodynamic, left ventricular reverse remodelling, sST2, 6MWT) at 3 months and 6 months post-aortic valve replacement.

It is expected that aortic valve replacement using a single strip of autologous pericardium will have good valve hemodynamic outcome, yield left ventricular reverse remodelling, decrease sST2 level, show upgrade in 6MWT, and have shorter aortic cross clamp time so that it can be an alternative to aortic valve replacement using mechanical prosthetic valve that is less expensive and have good outcomes in patient with aortic stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 10 years old
* Patients with aortic valve stenosis with an indication of aortic valve replacement having low to moderate surgical risk (EuroScore II <5)
* The patient or guardian (the research subject's parent) agrees to follow the study

Exclusion Criteria:

* Patients who have previously underwent aortic valve replacement
* Patients with aortic stenosis due to bicuspid aortic valve
* Patients with autoimmune disease
* Patients with mixed connective tissue disease

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2017-04-20 (Actual); Primary Completion 2020-01-20 (Estimated); Study Completion 2020-04-20 (Estimated)

PRIMARY OUTCOMES:
Change in Left Ventricular End Diastolic Diameter | before surgery, 3 months and 6 months after surgery
  Left Ventricular End Diastolic Diameter in mili meters assessed by Trans-thoracic Echocardiography measurement on M-mode
Change in Left Ventricular End Systolic Diameter | before surgery, 3 months and 6 months after surgery
  Left Ventricular End Systolic Diameter in mili meters assessed by Trans-thoracic Echocardiography measurement on M-mode
Change in Ejection Fraction Percentage | before surgery, 3 months and 6 months after surgery
  Ejection Fraction Percentage assessed by Trans-thoracic Echocardiography with modified Simpson's volumetric method (BiPlane measurement: apical 4 chambers and apical 2 chambers)
Change in 6 Minute Walking Test Performance (meters) | before surgery, 3 months and 6 months after surgery
  Subjects will be asked to walk for six minutes on a given track then the distance achieved will be measured in meters
Change in 6 Minute Walking Test Performance (METs) | before surgery, 3 months and 6 months after surgery
  The result of distance in meters of the six minute walking test will be converted to VO2max by the given formula:
  (distance in meters x 0.03) + 3.98 = VO2max
  Then the VO2max will be converted to METs by given formula:
  VO2max : 3.5 = METs
Change in Soluble Suppression of Tumorigenicity-2 (sST2) Level | before surgery, 3 months and 6 months after surgery
  Level of soluble Suppression of Tumorigenicity-2 measured in nano gram per mili Liters (ng/mL) by quantitative sandwich enzyme immunoassay technique assessed with Quantikinine Elisa

SECONDARY OUTCOMES:
Coaptation Height of Aortic Valve Leaflet in mili meters | at the time of surgery
  Aortic Valve Coaptation height measured in mili meters by Trans-oesophageal Echocardiography on mid-oesophageal long axis view
Effective Height of Aortic Valve in mili meters | at the time of surgery
  Effective Height of Aortic Valve measured in mili meters from Aortic annulus to the highest point of Aortic Valve coaptation by Trans-oesophageal Echocardiography in mid-oesophageal long axis view
Aortic Jet Velocity Value in m/s | before surgery
  Aortic Jet Velocity value measured in meters per second (m/s) by Color Wave Doppler on Trans-thoracic Echocardiography
Mean Trans-aortic Pressure Gradient Value in mmHg | before surgery
  Mean Trans-aortic Pressure Gradient Value measured in mili meters Hydrargyrum (mmHg) with Bernoulli equation on Trans-thoracic Echocardiography
Aortic Stenosis Severity | before surgery
  Aortic Stenosis Severity classified as mild, moderate, and severe based on Recommendations from European Association of Echocardiography and American Society of Echocardiography (EAE/ASE)
Aortic Regurgitation Severity | before surgery
  Aortic Regurgitation Severity classified as mild, moderate, and severe based on Recommendations from American Society of Echocardiography
Number of Valve Replacement and/or Repair | at the time of surgery
  Number of valves being replaced and/or repaired
Aortic Cross Clamp Time in minute | at the time of surgery
  The time from Aortic Cross Clamp On to Cross Clamp Off
Surgery Time in minute | at the time of surgery
  The time from first incision to finished closing surgical wound
Cardiopulmonary Bypass Time in minute | at the time of surgery
  The time from begin Cardiopulmonary Bypass (CPB) On to CPB Off
Duration of Hospitalization | at the time of surgery
  Number of days of Hospitalization since admission date to discharge date

OTHER OUTCOMES:
Duration of Intensive Care Unit Stay | at the time of surgery
  Number of hours in the Intensive Care Unit since after the surgery until subject is transferred to hospital ward
Duration of Ventilator Use | at the time of surgery
  Number of hours of breathing assisted with ventilator since intubation until extubation

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Dilawar, doctor, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] d'Arcy JL, Prendergast BD, Chambers JB, Ray SG, Bridgewater B. Valvular heart disease: the next cardiac epidemic. Heart. 2011 Jan;97(2):91-3. doi: 10.1136/hrt.2010.205096. Epub 2010 Dec 13. No abstract available. PMID 21149862
- [Result] Coffey S, Cairns BJ, Iung B. The modern epidemiology of heart valve disease. Heart. 2016 Jan;102(1):75-85. doi: 10.1136/heartjnl-2014-307020. Epub 2015 Nov 5. No abstract available. PMID 26541169
- [Result] Osnabrugge RL, Mylotte D, Head SJ, Van Mieghem NM, Nkomo VT, LeReun CM, Bogers AJ, Piazza N, Kappetein AP. Aortic stenosis in the elderly: disease prevalence and number of candidates for transcatheter aortic valve replacement: a meta-analysis and modeling study. J Am Coll Cardiol. 2013 Sep 10;62(11):1002-12. doi: 10.1016/j.jacc.2013.05.015. Epub 2013 May 30. PMID 23727214
- [Result] Maganti K, Rigolin VH, Sarano ME, Bonow RO. Valvular heart disease: diagnosis and management. Mayo Clin Proc. 2010 May;85(5):483-500. doi: 10.4065/mcp.2009.0706. PMID 20435842